CLINICAL TRIAL: NCT01140906
Title: A Randomised, Double-blind, Parallel-group, Placebo-controlled, Duloxetine-referenced, Fixed-dose Study Evaluating the Efficacy and Safety of Lu AA21004 (15 and 20 mg/Day) in the Acute Treatment of Adult Patients With Major Depressive Disorder
Brief Title: Randomised Placebo-controlled Duloxetine-referenced Study of Efficacy and Safety of 15 and 20 mg of Vortioxetine (Lu AA21004) in Acute Treatment of Major Depressive Disorder in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13267A; 2009-017523-26 (EudraCT Number)
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Placebo-controlled; Active reference; Multicenter study; Randomised study; Acute treatment
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vortioxetine: 15 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Vortioxetine: 20 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Duloxetine: 60 mg (Other): Active Reference
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Placebo — capsules, daily, orally
  Arms: Placebo
Drug: Vortioxetine (Lu AA21004) — encapsulated tablets, daily, orally
  Other Names: Brintellix
  Arms: Vortioxetine: 15 mg; Vortioxetine: 20 mg
Drug: Duloxetine — encapsulated capsules, daily, orally
  Other Names: Cymbalta®
  Arms: Duloxetine: 60 mg

SUMMARY:
The purpose of the study is to evaluate the efficacy, tolerability and the safety of two fixed doses of vortioxetine in the treatment of major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* The patient has recurrent MDD as the primary diagnosis according to DSM-IV-TR™ criteria (classification code 296.3x)
* The patient has a MADRS total score >=26
* The patient has a CGI-S score >=4
* The patient has had the current episode of MDE for >3 months

Exclusion Criteria:

* Any current anxiety psychiatric disorder as defined in the DSM-IV TR
* Current diagnosis or history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV TR
* Current diagnosis or history of alcohol or other substance abuse or dependence (excluding nicotine or caffeine) as defined in the DSM-IV TR
* Use of any psychoactive medication 2 weeks prior to screening and during the study
* The patient is at significant risk of suicide or has a score >=5 on Item 10 (suicidal thoughts) of the MADRS, or has attempted suicide within 6 months prior to the Screening Visit

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Derived] Adair M, Christensen MC, Florea I, Loft H, Fagiolini A. Vortioxetine in patients with major depressive disorder and high levels of anxiety symptoms: An updated analysis of efficacy and tolerability. J Affect Disord. 2023 May 1;328:345-354. doi: 10.1016/j.jad.2023.01.074. Epub 2023 Jan 26. PMID 36708956
- [Derived] Belzeaux R, Gorgievski V, Fiori LM, Lopez JP, Grenier J, Lin R, Nagy C, Ibrahim EC, Gascon E, Courtet P, Richard-Devantoy S, Berlim M, Chachamovich E, Theroux JF, Dumas S, Giros B, Rotzinger S, Soares CN, Foster JA, Mechawar N, Tall GG, Tzavara ET, Kennedy SH, Turecki G. GPR56/ADGRG1 is associated with response to antidepressant treatment. Nat Commun. 2020 Apr 2;11(1):1635. doi: 10.1038/s41467-020-15423-5. PMID 32242018
- [Derived] Christensen MC, Florea I, Loft H, McIntyre RS. Efficacy of vortioxetine in patients with major depressive disorder reporting childhood or recent trauma. J Affect Disord. 2020 Feb 15;263:258-266. doi: 10.1016/j.jad.2019.11.074. Epub 2019 Nov 13. PMID 31818787
- [Derived] Belzeaux R, Fiori LM, Lopez JP, Boucekine M, Boyer L, Blier P, Farzan F, Frey BN, Giacobbe P, Lam RW, Leri F, MacQueen GM, Milev R, Muller DJ, Parikh SV, Rotzinger S, Soares CN, Uher R, Foster JA, Kennedy SH, Turecki G. Predicting Worsening Suicidal Ideation With Clinical Features and Peripheral Expression of Messenger RNA and MicroRNA During Antidepressant Treatment. J Clin Psychiatry. 2019 May 7;80(3):18m12556. doi: 10.4088/JCP.18m12556. PMID 31087825
- [Derived] McIntyre RS, Florea I, Tonnoir B, Loft H, Lam RW, Christensen MC. Efficacy of Vortioxetine on Cognitive Functioning in Working Patients With Major Depressive Disorder. J Clin Psychiatry. 2017 Jan;78(1):115-121. doi: 10.4088/JCP.16m10744. PMID 27780334
- [Derived] Boulenger JP, Loft H, Olsen CK. Efficacy and safety of vortioxetine (Lu AA21004), 15 and 20 mg/day: a randomized, double-blind, placebo-controlled, duloxetine-referenced study in the acute treatment of adult patients with major depressive disorder. Int Clin Psychopharmacol. 2014 May;29(3):138-49. doi: 10.1097/YIC.0000000000000018. PMID 24257717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were selected from psychiatric settings (private practices), outpatient clinics, and inpatient hospitals.
Pre-assignment Details: At the Baseline Visit, patients who fulfilled the selection criteria were assigned to treatment with either placebo, vortioxetine 15 or 20 mg/day, or duloxetine 60 mg/day in a 1:1:1:1 ratio.
Groups:
- Vortioxetine 15 mg; Vortioxetine 20 mg: encapsulated tablets, daily, orally
- Duloxetine 60 mg: encapsulated capsules, daily, orally
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg
Started | 158 | 151 | 151 | 147
Completed | 133 | 117 | 125 | 131
Not Completed | 25 | 34 | 26 | 16
Not completed — Adverse Event | 7 | 10 | 17 | 7
Not completed — Lack of Efficacy | 6 | 8 | 2 | 1
Not completed — Non-compliance | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 5 | 3 | 2 | 1
Not completed — Withdrawal of consent | 6 | 6 | 2 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2
Not completed — Administrative or other reason | 0 | 5 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg | Total
Number analyzed (Participants) | 158 | 151 | 151 | 147 | 607
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (13.1) | 47.0 (14.6) | 46.2 (13.4) | 45.6 (13.6) | 46.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 97 | 91 | 102 | 400
  Male | 48 | 54 | 60 | 45 | 207
MADRS baseline total score [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. 9 of the items are based on patient report, and 1 is based on the rater's observation of the patients. Total score from 0 to 60. The higher the score, the more severe.
  units on a scale | 31.5 (3.6) | 31.8 (3.4) | 31.2 (3.4) | 31.2 (3.5) | 31.4 (3.5)
CGI-S baseline severity score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
  units on a scale | 4.9 (0.7) | 4.9 (0.6) | 4.8 (0.7) | 4.8 (0.7) | 4.8 (0.7)
HAM-A baseline total score [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
  units on a scale | 20.8 (6.6) | 21.3 (6.8) | 20.4 (6.9) | 20.5 (6.7) | 20.8 (6.7)
SDS total baseline score [Mean (Standard Deviation); unit: units on a scale] — The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe.
  units on a scale | 19.8 (6.0) | 20.6 (5.3) | 20.7 (4.8) | 20.5 (4.4) | 20.4 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MADRS Total Score After 8 Weeks of Treatment.
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
Time Frame: Baseline and Week 8
Population: Full-analysis set (FAS), mixed model for repeated measurements (MMRM)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg
Number analyzed (Participants) | 158 | 149 | 151 | 146
units on a scale | -11.70 (0.76) | -17.23 (0.79) | -18.79 (0.78) | -21.15 (0.77)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 15 mg; As soon as an endpoint was non-significant at the 0.025 level of significance, the testing procedure was stopped for all subsequent endpoints; Test type: Superiority or Other; p < 0.0001, MMRM — Since p-value <0.025, hierarchically testing continued; Mean Difference (Final Values) = -5.53, 95% CI 2-sided [-7.66 to -3.40], Standard Error of Mean 1.09 — To adjust for multiplicity the two doses of vortioxetine were tested separately versus placebo in the primary and key secondary efficacy analyses at a Bonferroni-corrected significance level of 0.025
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, MMRM — Since p-value <0.025, hierarchically testing continued; Mean Difference (Final Values) = -7.09, 95% CI 2-sided [-9.21 to -4.97], Standard Error of Mean 1.08 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p < 0.0001, MMRM — This treatment arm was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = -9.45, 95% CI 2-sided [-11.55 to -7.35], Standard Error of Mean 1.07

2. Secondary Outcome: Proportion of Responders at Week 8 (Response Defined as a >=50% Decrease in the MADRS Total Score From Baseline)
Time Frame: Week 8
Population: FAS, last observation carried forward (LOCF), Logistic Regression
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg
Number analyzed (Participants) | 158 | 149 | 151 | 146
percentage of patients | 32 | 57 | 62 | 74
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Adjusted Odds Ratio — Wald's test. Since p-value <0.025, hierarchically testing continued; Odds Ratio (OR) = 2.80, 95% CI 2-sided [1.76 to 4.47] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Adjusted Odds Ratio — Wald's test. Since p-value <0.025, hierarchically testing continued; Odds Ratio (OR) = 3.36, 95% CI 2-sided [2.10 to 5.36] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p < 0.0001, Adjusted Odds Ratio — This treatment arm was not in the testing sequence. A nominal p-value is provided; Odds Ratio (OR) = 5.94, 95% CI 2-sided [3.61 to 9.78]

3. Secondary Outcome: Change in Clinical Status Using CGI-I Score at Week 8
Description: The Clinical Global Impression - Global Improvement (CGI-I) is a 7-point scale rated from 1 (very much improved) to 7 (very much worse). The investigator rated the patient's overall improvement relative to baseline, whether or not, in the opinion of the investigator, this was entirely due to the drug treatment.
Time Frame: Week 8
Population: FAS, MMRM
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg
Number analyzed (Participants) | 158 | 149 | 151 | 146
units on a scale | 2.86 (0.09) | 2.18 (0.09) | 1.92 (0.09) | 1.75 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, MMRM — Since p-value <0.025, hierarchically testing continued; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-0.94 to -0.44], Standard Error of Mean 0.13 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, MMRM — Since p-value <0.025, hierarchically testing continued; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.20 to -0.70], Standard Error of Mean 0.13 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p < 0.0001, MMRM — This treatment arm was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-1.36 to -0.87], Standard Error of Mean 0.13

4. Secondary Outcome: Change From Baseline in MADRS Total Score After 8 Weeks of Treatment in Patients With Baseline HAM-A Total Score ≥20
Time Frame: Baseline and Week 8
Population: FAS, MMRM
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg
Number analyzed (Participants) | 89 | 87 | 80 | 80
units on a scale | -12.20 (1.09) | -17.44 (1.08) | -18.62 (1.15) | -20.91 (1.10)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0007, MMRM — Since p-value <0.025, hierarchically testing continued; Mean Difference (Final Values) = -5.24, 95% CI 2-sided [-8.25 to -2.22], Standard Error of Mean 1.53 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, MMRM — Since p-value <0.025, hierarchically testing continued; Mean Difference (Final Values) = -6.42, 95% CI 2-sided [-9.53 to -3.31], Standard Error of Mean 1.58 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p < 0.0001, MMRM — This treatment arm was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = -8.71, 95% CI 2-sided [-11.73 to -5.69], Standard Error of Mean 1.54

5. Secondary Outcome: Proportion of Remitters at Week 8 (Remission Defined as a MADRS Total Score <=10)
Time Frame: Week 8
Population: FAS, LOCF, Logistic Regression
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg
Number analyzed (Participants) | 158 | 149 | 151 | 146
percentage of patients | 19 | 35 | 38 | 54
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0016, Adjusted Odds Ratio — Wald's test. Since p-value <0.025, hierarchically testing continued; Odds Ratio (OR) = 2.32, 95% CI 2-sided [1.37 to 3.91] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, Adjusted Odds Ratio — Wald's test. Since p-value <0.025, hierarchically testing continued; Odds Ratio (OR) = 2.65, 95% CI 2-sided [1.58 to 4.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p < 0.0001, Adjusted for Odds Ratio — Wald's test. This treatment arm was not in the testing sequence. A nominal p-value is provided; Odds Ratio (OR) = 5.01, 95% CI 2-sided [2.99 to 8.37]

6. Secondary Outcome: Change From Baseline in SDS Total Score After 8 Weeks of Treatment
Description: The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe.
Time Frame: Baseline and Week 8
Population: FAS, MMRM
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg
Number analyzed (Participants) | 115 | 97 | 107 | 99
units on a scale | -4.46 (0.82) | -7.70 (0.89) | -8.38 (0.85) | -11.39 (0.85)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 15 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0054, MMRM — Since p-value <0.025, hierarchically testing continued; Mean Difference (Final Values) = -3.24, 95% CI 2-sided [-5.51 to -0.97], Standard Error of Mean 1.16 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0005, MMRM — Since p-value <0.025, hierarchically testing continued; Mean Difference (Final Values) = -3.92, 95% CI 2-sided [-6.11 to -1.73], Standard Error of Mean 1.11 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p < 0.0001, MMRM — This treatment arm was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = -6.93, 95% CI 2-sided [-9.16 to -4.70], Standard Error of Mean 1.13

7. Secondary Outcome: Change From Baseline in ASEX Total Score After 8 Weeks of Treatment
Description: The Arizona Sexual Experience Scale (ASEX) is a 5-item, patient self-rated scale that evaluates a patient's recent sexual experience. Patients are asked to assess their own experience over the last week (for example, "How strong is your sex drive?", "Are your orgasms satisfying?") and respond on a 6-point scale for each item. The ASEX is used to identify individuals with sexual dysfunction. Possible total score ranges from 5 to 30, with the higher score indicating more patient sexual dysfunction. A negative change indicates a lower sexual dysfunction.
Time Frame: Baseline and Week 8
Population: FAS, MMRM
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg
Number analyzed (Participants) | 156 | 147 | 148 | 144
units on a scale | 0.28 (0.42) | -0.39 (0.43) | -0.20 (0.43) | -1.25 (0.42)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 15 mg; Test type: Superiority or Other; p = 0.2524, MMRM — A nominal p-value is provided; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.83 to 0.48], Standard Error of Mean 0.59 — No correction for multiplicity was made
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p = 0.4186, MMRM — A nominal p-value is provided; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.64 to 0.68], Standard Error of Mean 0.59 — No correction for multiplicity was made

8. Secondary Outcome: Potential Discontinuation Symptoms After Abrupt Discontinuation of Treatment With Vortioxetine
Description: The Discontinuation-Emergent Signs and Symptoms Scale (DESS) was designed to evaluate possible effects of discontinuation of antidepressant therapy. It is a clinician-rated instrument that queries for signs and symptoms on a 43-item checklist (for example, agitation, insomnia, fatigue, and dizziness) to assess whether the item (event) is discontinuation-emergent. A new or worsened event reported after discontinuation of therapy scores 1 point on the checklist, and the DESS total score is the sum of all positive scores on the checklist. A higher score indicates more symptoms.
Time Frame: Change from Week 8 in DESS total score analyzed at Week 10
Population: All Patients Completed Set (APCS), OC, Analysis of Covariance (ANCOVA)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg
Number analyzed (Participants) | 121 | 116 | 120 | 127
units on a scale | 0.15 (0.30) | 0.01 (0.31) | 0.72 (0.31) | 2.28 (0.30)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 15 mg; Test type: Superiority or Other; p = 0.7372, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.95 to 0.67], Standard Error of Mean 0.41
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p = 0.1690, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-0.24 to 1.37], Standard Error of Mean 0.41

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 8-week double-blind treatment period and 4-week safety follow-up period Other Adverse Events: 8-week double-blind treatment period
Arm/Group | Placebo | Vortioxetine 15 mg | Vortioxetine 20 mg | Duloxetine 60 mg
Serious Adverse Events (participants affected / at risk) | 0/158 | 0/151 | 2/151 | 3/147
Other Adverse Events (participants affected / at risk) | 44/158 | 61/151 | 70/151 | 67/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=158) | Vortioxetine 15 mg (N=151) | Vortioxetine 20 mg (N=151) | Duloxetine 60 mg (N=147)
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 1 | 0
Self injurious behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/110 | 0/97 | 0/91 | 1/102
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=158) | Vortioxetine 15 mg (N=151) | Vortioxetine 20 mg (N=151) | Duloxetine 60 mg (N=147)
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 11 | 9
Dry mouth (Gastrointestinal disorders) | 5 | 5 | 9 | 14
Nausea (Gastrointestinal disorders) | 16 | 40 | 48 | 45
Fatigue (General disorders) | 4 | 6 | 5 | 8
Dizziness (Nervous system disorders) | 10 | 7 | 7 | 15
Headache (Nervous system disorders) | 12 | 16 | 19 | 16
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 5 | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study will be published at the discretion of H. Lundbeck A/S. H. Lundbeck A/S will ensure that the authorship of all publications based on this study is in accordance with the criteria defined by the International Committee of Medical Journal Editors (ICMJE).

The primary publication must be published before any secondary publications.